CLINICAL TRIAL: NCT00728637
Title: Effectiveness of a Family Heart Health Intervention Trial (FIT Heart I)
Brief Title: Evaluating the Effectiveness of a Family Heart Health Educational Program (The FIT-Heart Study)
Acronym: FIT-Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lori Mosca, Professor of Medicine, Columbia University., Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAA5856; R01HL075101 (NIH)
Record Dates: First submitted 2008-08-04; First posted 2008-08-06 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
Keywords: Prevention
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants took part in the Family Passport to Heart Health Program.
  Interventions: Behavioral: Family Passport to Heart Health Program
- 2 (Active Comparator): Participants took part in a control group.
  Interventions: Behavioral: General Educational Materials

INTERVENTIONS:
Behavioral: Family Passport to Heart Health Program — Participants in this group received personalized heart disease risk factor screening at the baseline study visit. They were taught lifestyle approaches to risk reduction based upon national heart disease prevention guidelines, including the Adult Treatment Panel (ATP) III recommendations for improving blood cholesterol levels with a TLC diet. Participants had regular contact with study staff and will receive individualized feedback throughout the study.
  Arms: 1
Behavioral: General Educational Materials — Participants in the control group received an educational brochure about heart health at the baseline study visit.
  Arms: 2

SUMMARY:
The primary objective of the FIT Heart Study was to test the effectiveness of a hospital-based standardized screening and educational intervention targeted to family members of patients hospitalized with CVD, to increase adherence to CVD prevention guidelines.

DETAILED DESCRIPTION:
FIT Heart was a randomized controlled trial that tested a novel systems approach to increase adherence to national prevention guidelines among family members of patients hospitalized with CVD. Participants were blood relatives or cohabitants of patients hospitalized with atherosclerotic cardiovascular disease, aged 20-79 years, did not have established cardiovascular disease or diabetes, and spoke English or Spanish. Participants randomized to a special intervention group received behavioral counseling and education on diet and physical activity; personalized risk factor screening and immediate feedback; and reinforcement and follow-up throughout the year. The control group received a brief CVD prevention message in the form of a handout. All participants received standardized assessments of diet, lifestyle, and CVD risk factors at baseline and 1 year (94% follow-up). The main findings have been published showing the mean percent change in LDL-cholesterol level from baseline to 1-year improved in both groups and was not significantly different in the special intervention vs. control group (-1% vs. -2%; p=.64).

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 5 years after study entry
* Willing to return at Year 1 for a repeat study evaluation
* Family member was hospitalized with acute atherosclerotic cardiovascular disease, including catheter-based procedures and coronary artery bypass grafting
* Speaks either English or Spanish

Exclusion Criteria:

* Established cardiovascular disease, diabetes, active liver disease, or long-term kidney disease
* Life expectancy less than 5 years from study entry
* Prescription of a special diet that is not compatible with the TLC diet
* Participation in a clinical drug study in the 3 months before study entry
* Pregnant or planning to become pregnant

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean percent reduction in low-density lipoprotein (LDL) cholesterol levels in the special intervention group versus the control group | Measured at Year 1

SECONDARY OUTCOMES:
Mean percent change in high density lipoprotein (HDL) cholesterol levels in the special intervention group versus the control group | Measured at Year 1
Attainment of the Therapeutic Lifestyle Change (TLC) diet | Measured at Year 1
Change in lipoproteins, high sensitivity C-reactive protein (hsCRP), blood pressure, body mass index, waist circumference, Framingham risk, and diet score in the special intervention group versus the control group | Measured at Year 1
Cost effectiveness of the personalized educational program to reduce LDL cholesterol levels and cost per life saved | Measured at Year 1
Impact of hsCRP beyond traditional risk factors on attainment of prevention goals | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Lori Mosca, MD, MPH, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Edelman DJ, Gao Q, Mosca L. Predictors and barriers to timely medical follow-up after cardiovascular disease risk factor screening according to race/ethnicity. J Natl Med Assoc. 2008 May;100(5):534-9. doi: 10.1016/s0027-9684(15)31299-2. PMID 18507205
- [Result] Mochari H, Gao Q, Mosca L. Validation of the MEDFICTS dietary assessment questionnaire in a diverse population. J Am Diet Assoc. 2008 May;108(5):817-22. doi: 10.1016/j.jada.2008.02.021. PMID 18442505
- [Result] Fischer Aggarwal BA, Liao M, Mosca L. Physical activity as a potential mechanism through which social support may reduce cardiovascular disease risk. J Cardiovasc Nurs. 2008 Mar-Apr;23(2):90-6. doi: 10.1097/01.JCN.0000305074.43775.d8. PMID 18382248
- [Result] Aggarwal B, Liao M, Mosca L. Predictors of physical activity at 1 year in a randomized controlled trial of family members of patients with cardiovascular disease. J Cardiovasc Nurs. 2010 Nov-Dec;25(6):444-9. doi: 10.1097/JCN.0b013e3181defd3e. PMID 20856131
- [Result] Aggarwal B, Liao M, Allegrante JP, Mosca L. Low social support level is associated with non-adherence to diet at 1 year in the Family Intervention Trial for Heart Health (FIT Heart). J Nutr Educ Behav. 2010 Nov-Dec;42(6):380-8. doi: 10.1016/j.jneb.2009.08.006. Epub 2010 Aug 8. PMID 20696617
- [Result] Mosca L, Mochari H, Liao M, Christian AH, Edelman DJ, Aggarwal B, Oz MC. A novel family-based intervention trial to improve heart health: FIT Heart: results of a randomized controlled trial. Circ Cardiovasc Qual Outcomes. 2008 Nov;1(2):98-106. doi: 10.1161/CIRCOUTCOMES.108.825786. Epub 2008 Nov 12. PMID 20031796
- [Result] Aggarwal B, Liao M, Christian A, Mosca L. Influence of caregiving on lifestyle and psychosocial risk factors among family members of patients hospitalized with cardiovascular disease. J Gen Intern Med. 2009 Jan;24(1):93-8. doi: 10.1007/s11606-008-0852-1. Epub 2008 Nov 8. PMID 18998190
- [Result] Mochari-Greenberger H, Mosca L. Caregiver burden and nonachievement of healthy lifestyle behaviors among family caregivers of cardiovascular disease patients. Am J Health Promot. 2012 Nov-Dec;27(2):84-9. doi: 10.4278/ajhp.110606-QUAN-241. PMID 23113777
- [Result] Mochari-Greenberger H, Terry MB, Mosca L. Sex, age, and race/ethnicity do not modify the effectiveness of a diet intervention among family members of hospitalized cardiovascular disease patients. J Nutr Educ Behav. 2011 Sep-Oct;43(5):366-73. doi: 10.1016/j.jneb.2011.01.014. PMID 21906549
- [Result] Mochari-Greenberger H, Terry MB, Mosca L. Does stage of change modify the effectiveness of an educational intervention to improve diet among family members of hospitalized cardiovascular disease patients? J Am Diet Assoc. 2010 Jul;110(7):1027-35. doi: 10.1016/j.jada.2010.04.012. PMID 20630159
- [Result] Parikh P, Mochari H, Mosca L. Clinical utility of a fingerstick technology to identify individuals with abnormal blood lipids and high-sensitivity C-reactive protein levels. Am J Health Promot. 2009 Mar-Apr;23(4):279-82. doi: 10.4278/ajhp.071221140. PMID 19288850
- [Result] Mochari H, Grbic JT, Mosca L. Usefulness of self-reported periodontal disease to identify individuals with elevated inflammatory markers at risk of cardiovascular disease. Am J Cardiol. 2008 Dec 1;102(11):1509-13. doi: 10.1016/j.amjcard.2008.07.047. Epub 2008 Sep 15. PMID 19026305
- [Result] Nawathe AC, Glied SA, Weintraub WS, Mosca LJ. The effect of a cardiovascular educational intervention on healthcare utilization and costs. Am J Manag Care. 2010 May;16(5):339-46. PMID 20469954